CLINICAL TRIAL: NCT01563133
Title: Clinical Evaluation Of NCLE in The Lymph Nodes Along With Masses and Cystic Tumors of the Pancreas
Brief Title: Clinical Evaluation Of Needle-based Confocal Laser Endomicroscopy in The Lymph Nodes Along With Masses and Cystic Tumors of the Pancreas
Acronym: CONTACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mauna Kea Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MKT-2012-nCLE-02
Record Dates: First submitted 2012-03-22; First posted 2012-03-26 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic Adenoma; Pancreatic Cancer; Pancreatic Islet Cell Tumors; Lymph Node; Lymphadenopathy
Keywords: endomicroscopy; needle-based; pancreatic; cyst; mass; EUSFNA
MeSH Terms: conditions — Pancreatic Cyst; Pancreatic Neoplasms; Pancreatic adenoma; Adenoma, Islet Cell; Lymphadenopathy; Cysts; Arachnodactyly | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lymph nodes, pancreatic masses & cysts (Other)
  Interventions: Procedure: EUS-FNA; Device: nCLE

INTERVENTIONS:
Procedure: EUS-FNA — Endoscopic ultrasound fine needle aspiration: ultrasound endoscopy of a lesion with aspiration of the lesion fluid through a needle
  Other Names: ultrasonographic endoscopy; EUS-guided FNA
Device: nCLE — needle-based Confocal Laser Endomicroscopy

SUMMARY:
This study focuses on three different lesions: pancreatic cysts, lymph nodes near the gastrointestinal tract and pancreatic masses.

On one hand, the results obtained during previous studies are more advanced for the assessment of the diagnostic performance of Cellvizio needle-based Confocal Laser Endomicroscopy (nCLE) system for Pancreatic cysts. Safety and technical feasibility have already been performed, and an interpretation criteria classification exists. On the other hand, results for pancreatic masses and Lymph nodes are less developed.

The study therefore comprises two sub-studies, one on the pancreatic cysts, and another on pancreatic masses and lymph nodes.

1. Cysts The primary hypothesis of the study is that using nCLE in addition to EUS-FNA and tissue sampling allows better characterization of pancreatic cysts and improves appropriate therapeutic decision-making.

   For physicians, integrating nCLE into the diagnostic algorithm of pancreatic cysts could impact patient management by :
   * Ruling out malignancy for patients with benign appearing nCLE images.
   * Characterizing more malignant tumors in the pancreas.
2. Pancreatic masses and Lymph nodes The primary hypothesis of the study is that in vivo imaging of lymph-nodes near the gastrointestinal tract and pancreatic masses during EUS-FNA procedures is feasible and that descriptive criteria can be defined to further differentiate the different types of lesions.

DETAILED DESCRIPTION:
1. Medical background Pancreatic cancer is the fourth leading cause of cancer-related death in the United States. This disease is associated with a high mortality rate: the 5-year survival rate is estimated to be 4%. This is mainly due to the fact that the disease is often discovered at an already advanced disease state, which carries a dismal prognosis.

   1.1. Pancreatic Cysts

   Pancreatic cysts are quite rare, but are being increasingly recognized due to the expanding use of cross-sectional imaging. They are classified into three main classes:
   * Pseudocysts
   * Serous cysts : either serous cystic neoplasms (SCN) or Solid pseudo-papillary neoplasm (SPN)
   * Mucinous cystic neoplasms : either Intraductal Papillary Mucinous Neoplasm (IPMN) or mucinous cystadenomas/mucinous cystadenocarcinoma(MCN) Mucinous cystic neoplasms are considered to be malignant or pre-malignant and are considered for surgical resection, whereas pseudocysts and serous cysts are considered benign and with a low potential for malignancy. Pseudocysts and serous cysts are usually only considered for surgical resection when symptomatic or enlarging.

   1.2. Pancreatic masses Pancreatic solid masses can be either exocrine or endocrine tumors, or metastatic.Exocrine tumors are by far the most common type of pancreas cancer. Most of them are malignant. About 96% of cancers of the exocrine pancreas are adenocarcinomas, which is the most aggressive form of pancreas cancer.Endocrine tumors are uncommon. They represent 4% of pancreas tumors. They are known as neuroendocrine tumors (NETs), or islet cell tumors. These tumors can be benign or malignant.

   1.3. Lymph nodes Lymph nodes are examined in a patient with a suspicion of, or confirmed, cancer, as part of the staging. They may be either normal, inflammatory, or malignant.
2. Clinical background

   2.1. EUSFNA Endoscopic Ultrasound (EUS) is the diagnostic method of choice when a pancreatic lesion is found incidentally on cross-sectional imaging. Endoscopic UltraSound-guided Fine Needle Aspiration (EUS FNA) (respectively Endobronchial Ultrasound-guided Fine Needle Aspiration (EBUS FNA)) are procedures where a target tissue in proximity to the GI tract (respectively the pulmonary tract) is biopsied using a fine needle guided in real time by an ultrasound probe fixed at the tip of an endoscope.It may therefore be applied to pancreatic lesions, or lymph nodes examination.

   2.2. nCLE The principle of needle-based Confocal Laser Endomicroscopy (nCLE) is to image organs within or adjacent to the GI or respiratory tracts with a miniprobe inserted through an endoscopic needle. The fundamental technology as well as the principle of operation of nCLE are substantially similar to pCLE.
3. Clinical evidence More than 100 patients have already underwent an nCLE procedure, in the past studies. A first feasibility study enabled to define the final type of probe which would fit into a EUSFNA needle, and the INSPECT study enabled to define interpretation criteria on the micro-structure of pancreatic cysts. Less data is available on pancreatic masses and lymph nodes, except for a few images done in the first feasibility study.
4. Objectives

   4.1. Cysts 4.1.1. The primary objective of the study is to assess the diagnostic performance of the Cellvizio nCLE system in diagnosing pancreatic cysts, when associated with other diagnostic information.

   4.1.2. The secondary objectives are to assess the potential impact of the Cellvizio nCLE system on patient management and validate the interpretation classification criteria that were created during the previous INSPECT study on cysts.

   4.2. Pancreatic masses and Lymph nodes 4.2.1. The primary objective of the study is to define criteria of nCLE sequences in lymph nodes and pancreatic masses.

   4.2.2. The secondary objectives are to evaluate feasibility and safety of the Cellvizio nCLE during EUS-FNA procedures, build an atlas of images of nCLE sequences of pancreatic masses and lymph nodes, and, finally, retrospectively assess the diagnostic performance of nCLE in the diagnosis of pancreatic masses and lymph nodes, when associated with other diagnostic information
5. Design This study will be conducted in three centers in France.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years of age.
* Patient indicated for a first EUS-FNA for a pancreatic cyst, lymph node or pancreatic mass, or
* Patients who had previous non-diagnostic tissue sampling taken during a previous EUS-FNA for pancreatic cyst, lymph nodes, pancreatic mass, more than three months ago.
* Patient with known pancreatic cyst or mass detected at cross-sectional imaging or suspicious lymph nodes reachable via EUSFNA
* Willing and able to comply with study procedures and provide written informed consent to participate in the study.

Add for lymph nodes:

- any lymph node reachable with EUS-FNA

Add for pancreatic mass:

* any size
* any location in the pancreas

Exclusion Criteria:

* Subjects for whom EUS-FNA procedures are contraindicated
* Known allergy to fluorescein dye
* If female, pregnant based on a positive hCG serum or an in vitro diagnostic test result or breast-feeding

Add for cysts:

* Subject with multiple cysts
* size < 20mm in diameter
* previous EUS-FNA procedure performed less than 3 months ago - Patients suffering chronic calcifying pancreatitis

Add for lymph nodes:

* size < 5mm in diameter
* If patients present several suspicious lymph nodes, only one of them will be imaged during the nCLE procedure

Add for pancreatic mass:

- If patient present several pancreatic masses, only one of them will be imaged during the nCLE procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2012-06; Primary Completion 2016-03-02 (Actual); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of the Cellvizio nCLE system in the characterization of pancreatic cysts | Within 6 months after the end of Follow-up period
Descriptive criteria in nCLE sequences for the characterization of pancreatic masses and lymph nodes | Within one year after the end of the follow-up period

SECONDARY OUTCOMES:
Impact of the Cellvizio nCLE system on the management of a patient with pancreatic cyst | Within one year after the end of the follow-up period
Validation of the interpretation criteria classification for pancreatic cysts | within 6 months after the end of the follow-up period
Atlas of images of nCLE sequences of pancreatic masses and lymph nodes during EUS-FNA | within 3 months of the end of the follow-up period
Diagnostic performance of nCLE in the diagnosis of pancreatic masses and lymph nodes, when associated with other diagnostic information | within one year after the end of the follow-up period
Feasibility and safety data on nCLE during EUS-FNA procedure | Within 3 months after the end of the enrollment period

CONTACTS AND LOCATIONS:
Overall Officials: Marc Giovannini, MD, Principal Investigator — Institut Paoli-Calmettes
Locations (3):
- France (3):
  - Hôpital Saint-Philibert, Lomme
  - Hôpital Jean Mermoz, Lyon
  - Institut Paoli Calmettes, Marseille

REFERENCES:
- [Background] Adsay NV. Cystic neoplasia of the pancreas: pathology and biology. J Gastrointest Surg. 2008 Mar;12(3):401-4. doi: 10.1007/s11605-007-0348-z. Epub 2007 Oct 24. PMID 17957438
- [Background] Levy MJ, Clain JE. Evaluation and management of cystic pancreatic tumors: emphasis on the role of EUS FNA. Clin Gastroenterol Hepatol. 2004 Aug;2(8):639-53. doi: 10.1016/s1542-3565(04)00235-6. PMID 15290655
- [Background] Hutchins GF, Draganov PV. Cystic neoplasms of the pancreas: a diagnostic challenge. World J Gastroenterol. 2009 Jan 7;15(1):48-54. doi: 10.3748/wjg.15.48. PMID 19115467
- [Background] Attasaranya S, Pais S, LeBlanc J, McHenry L, Sherman S, DeWitt JM. Endoscopic ultrasound-guided fine needle aspiration and cyst fluid analysis for pancreatic cysts. JOP. 2007 Sep 7;8(5):553-63. PMID 17873459
- [Background] Becker V, Vercauteren T, von Weyhern CH, Prinz C, Schmid RM, Meining A. High-resolution miniprobe-based confocal microscopy in combination with video mosaicing (with video). Gastrointest Endosc. 2007 Nov;66(5):1001-7. doi: 10.1016/j.gie.2007.04.015. Epub 2007 Sep 4. PMID 17767932
- [Background] Meining A, Saur D, Bajbouj M, Becker V, Peltier E, Hofler H, von Weyhern CH, Schmid RM, Prinz C. In vivo histopathology for detection of gastrointestinal neoplasia with a portable, confocal miniprobe: an examiner blinded analysis. Clin Gastroenterol Hepatol. 2007 Nov;5(11):1261-7. doi: 10.1016/j.cgh.2007.05.019. Epub 2007 Aug 6. PMID 17689297
- [Background] Kiesslich R, Gossner L, Goetz M, Dahlmann A, Vieth M, Stolte M, Hoffman A, Jung M, Nafe B, Galle PR, Neurath MF. In vivo histology of Barrett's esophagus and associated neoplasia by confocal laser endomicroscopy. Clin Gastroenterol Hepatol. 2006 Aug;4(8):979-87. doi: 10.1016/j.cgh.2006.05.010. Epub 2006 Jul 13. PMID 16843068
- [Background] Pohl H, Rosch T, Vieth M, Koch M, Becker V, Anders M, Khalifa AC, Meining A. Miniprobe confocal laser microscopy for the detection of invisible neoplasia in patients with Barrett's oesophagus. Gut. 2008 Dec;57(12):1648-53. doi: 10.1136/gut.2008.157461. Epub 2008 Aug 28. PMID 18755886
- [Background] Buchner AM, Shahid MW, Heckman MG, Krishna M, Ghabril M, Hasan M, Crook JE, Gomez V, Raimondo M, Woodward T, Wolfsen HC, Wallace MB. Comparison of probe-based confocal laser endomicroscopy with virtual chromoendoscopy for classification of colon polyps. Gastroenterology. 2010 Mar;138(3):834-42. doi: 10.1053/j.gastro.2009.10.053. Epub 2009 Nov 10. PMID 19909747
- [Background] Meining A, Frimberger E, Becker V, Von Delius S, Von Weyhern CH, Schmid RM, Prinz C. Detection of cholangiocarcinoma in vivo using miniprobe-based confocal fluorescence microscopy. Clin Gastroenterol Hepatol. 2008 Sep;6(9):1057-60. doi: 10.1016/j.cgh.2008.04.014. Epub 2008 Jul 17. PMID 18639496
- [Background] Meining A, Phillip V, Gaa J, Prinz C, Schmid RM. Pancreaticoscopy with miniprobe-based confocal laser-scanning microscopy of an intraductal papillary mucinous neoplasm (with video). Gastrointest Endosc. 2009 May;69(6):1178-80. doi: 10.1016/j.gie.2008.06.013. Epub 2009 Jan 18. No abstract available. PMID 19152895
- [Background] Konda VJ, Aslanian HR, Wallace MB, Siddiqui UD, Hart J, Waxman I. First assessment of needle-based confocal laser endomicroscopy during EUS-FNA procedures of the pancreas (with videos). Gastrointest Endosc. 2011 Nov;74(5):1049-60. doi: 10.1016/j.gie.2011.07.018. Epub 2011 Sep 15. PMID 21924718
- [Background] Giovannini, M., Monges, G.M., Caillol,F., Bories, E., Pesenti C. Feasibility of Intra-Tumoral Confocal Microscopy Under EUS Guidance (EUS-CM)
- [Background] Wallace MB, Meining A, Canto MI, Fockens P, Miehlke S, Roesch T, Lightdale CJ, Pohl H, Carr-Locke D, Lohr M, Coron E, Filoche B, Giovannini M, Moreau J, Schmidt C, Kiesslich R. The safety of intravenous fluorescein for confocal laser endomicroscopy in the gastrointestinal tract. Aliment Pharmacol Ther. 2010 Mar;31(5):548-52. doi: 10.1111/j.1365-2036.2009.04207.x. Epub 2009 Nov 30. PMID 20002025
- [Background] Becker V, Wallace MB, Fockens P, von Delius S, Woodward TA, Raimondo M, Voermans RP, Meining A. Needle-based confocal endomicroscopy for in vivo histology of intra-abdominal organs: first results in a porcine model (with videos). Gastrointest Endosc. 2010 Jun;71(7):1260-6. doi: 10.1016/j.gie.2010.01.010. Epub 2010 Apr 24. PMID 20421104
- [Background] Khalid A, Brugge W. ACG practice guidelines for the diagnosis and management of neoplastic pancreatic cysts. Am J Gastroenterol. 2007 Oct;102(10):2339-49. doi: 10.1111/j.1572-0241.2007.01516.x. Epub 2007 Aug 31. PMID 17764489
- [Background] Bhutani MS. Role of endoscopic ultrasonography in the diagnosis and treatment of cystic tumors of the pancreas. JOP. 2004 Jul;5(4):266-72. PMID 15254361
- [Background] Sahani DV, Kadavigere R, Saokar A, Fernandez-del Castillo C, Brugge WR, Hahn PF. Cystic pancreatic lesions: a simple imaging-based classification system for guiding management. Radiographics. 2005 Nov-Dec;25(6):1471-84. doi: 10.1148/rg.256045161. PMID 16284129
- [Derived] Palazzo M, Sauvanet A, Gincul R, Borbath I, Vanbiervliet G, Bourdariat R, Lemaistre AI, Pujol B, Caillol F, Palazzo L, Aubert A, Maire F, Buscail L, Giovannini M, Marque S, Napoleon B. Impact of needle-based confocal laser endomicroscopy on the therapeutic management of single pancreatic cystic lesions. Surg Endosc. 2020 Jun;34(6):2532-2540. doi: 10.1007/s00464-019-07062-9. Epub 2019 Aug 13. PMID 31410626
- [Derived] Napoleon B, Palazzo M, Lemaistre AI, Caillol F, Palazzo L, Aubert A, Buscail L, Maire F, Morellon BM, Pujol B, Giovannini M. Needle-based confocal laser endomicroscopy of pancreatic cystic lesions: a prospective multicenter validation study in patients with definite diagnosis. Endoscopy. 2019 Sep;51(9):825-835. doi: 10.1055/a-0732-5356. Epub 2018 Oct 22. PMID 30347425
- [Derived] Giovannini M, Caillol F, Monges G, Poizat F, Lemaistre AI, Pujol B, Lucidarme D, Palazzo L, Napoleon B. Endoscopic ultrasound-guided needle-based confocal laser endomicroscopy in solid pancreatic masses. Endoscopy. 2016 Oct;48(10):892-8. doi: 10.1055/s-0042-112573. Epub 2016 Aug 30. PMID 27576181
- [Derived] Napoleon B, Lemaistre AI, Pujol B, Caillol F, Lucidarme D, Bourdariat R, Morellon-Mialhe B, Fumex F, Lefort C, Lepilliez V, Palazzo L, Monges G, Filoche B, Giovannini M. A novel approach to the diagnosis of pancreatic serous cystadenoma: needle-based confocal laser endomicroscopy. Endoscopy. 2015 Jan;47(1):26-32. doi: 10.1055/s-0034-1390693. Epub 2014 Oct 17. PMID 25325684